CLINICAL TRIAL: NCT02525094
Title: A Phase 2a, Randomized, Double-blinded, Placebo-controlled Study to Evaluate the Efficacy and Safety of MEDI9929 in Adult Subjects With Moderate-to-Severe Atopic Dermatitis
Brief Title: Phase 2a Study to Evaluate the Efficacy and Safety of MEDI9929 in Adults With Atopic Dermatitis
Acronym: ALLEVIAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5240C00001
Record Dates: First submitted 2015-07-29; First posted 2015-08-17 (Estimated); Results first posted 2018-02-15 (Actual); Last update posted 2018-02-15 (Actual); Status verified 2018-01

CONDITIONS: Atopic Dermatitis
Keywords: Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — tezepelumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MEDI9929 280 mg (Experimental): Participants will receive 6 subcutaneous doses of MEDI9929 280 mg every 2 weeks for 12 weeks, with the last dose at Week 10.
  Interventions: Biological: MEDI9929
- Placebo (Placebo Comparator): Participants will receive 6 subcutaneous doses of placebo every 2 weeks for 12 weeks, with the last dose at Week 10.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: MEDI9929 — Participants will receive 6 subcutaneous doses of MEDI9929 280 mg every 2 weeks for 12 weeks, with the last dose at Week 10.
  Arms: MEDI9929 280 mg
Biological: Placebo — Participants will receive 6 subcutaneous doses of placebo every 2 weeks for 12 weeks, with the last dose at Week 10.
  Arms: Placebo

SUMMARY:
To assess the efficacy and safety of MEDI9929 in adult subjects with Atopic Dermatitis

DETAILED DESCRIPTION:
This is a Phase 2a, randomized, double-blinded, placebo-controlled study to evaluate the efficacy and safety of MEDI9929 administered subcutaneously to adult subjects with moderate to severe Atopic Dermatitis. Subjects will be randomized in a 1:1 fashion and will be stratified at screening. Approximately 100 subjects are planned to be randomized at approximately 35 sites in 6 countries

ELIGIBILITY:
Inclusion Criteria:

* AD meeting Hanifin and Rajka criteria
* Age 18-75 years inclusive at screening
* Atopic dermatitis that affects greater than/equal to 10% body surface area
* Moderate to severe AD
* Effective birth control in line with protocol details

Exclusion Criteria:

* Active dermatologic conditions which may confuse the diagnosis of Atopic Dermatitis
* Hepatitis B, C or HIV
* Pregnant or breastfeeding
* History of anaphylaxis following any biologic therapy
* History of clinically significant infections within 4 weeks prior to Visit 3
* Diagnosis of helminth parasitic infection within 6 months to screening
* History of Cancer except basal cell
* Receipt of any marketed or investigational biologic agent within 4 months to visit 3
* Any clinically relevant abnormal finding
* Major surgery within 8 weeks prior to Visit 1

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2015-08-15 (Actual); Primary Completion 2016-05-09 (Actual); Study Completion 2016-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Simpson, MD, Principal Investigator — Oregon Health and Science University; Roderick Mcphee, MD, Study Director — MedImmune LLC
Locations (29):
- United States (8):
  - Research Site, North Miami Beach, Florida
  - Research Site, Tampa, Florida
  - Research Site, Arlington Hts, Illinois
  - Research Site, Carmel, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, Berlin, New Jersey
  - Research Site, Charlotte, North Carolina
  - Research Site, Portland, Oregon
- Australia (3):
  - Research Site, ACT
  - Research Site, Liverpool
  - Research Site, Woolloongabba
- Canada (3):
  - Research Site, Surrey, British Columbia
  - Research Site, Barrie, Ontario
  - Research Site, Québec, Quebec
- Germany (7):
  - Research Site, Berlin
  - Research Site, Frankfurt am Main
  - Research Site, Gera
  - Research Site, Hanover
  - Research Site, Leipzig
  - Research Site, München
  - Research Site, Münster
- Hungary (6):
  - Research Site, Debrecen
  - Research Site, Kaposvár
  - Research Site, Miskolc
  - Research Site, Pécs
  - Research Site, Szeged
  - Research Site, Szombathely
- New Zealand (2):
  - Research Site, Tauranga
  - Research Site, Wellington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 15Aug2015 to 15Jul2016.
Pre-assignment Details: A total of 155 participants were screened, of which 113 were randomized into the study.
Groups:
- Placebo: Participants received 6 subcutaneous doses of placebo every 2 weeks for 12 weeks (with the last dose at Week 10) and were followed up till Week 22. Additionally, the participants received maintenance therapy of Class 3 topical corticosteroids (TCS) cream or ointment for lesional skin from the start of the run-in period (Visit 2, Week -2) to Week 22.
- MEDI9929 280 mg: Participants received 6 subcutaneous doses of MEDI9929 280 mg every 2 weeks for 12 weeks (with the last dose at Week 10) and were followed up till Week 22. Additionally, the participants received maintenance therapy of Class 3 topical corticosteroids (TCS) cream or ointment for lesional skin from the start of the run-in period (Visit 2, Week -2) to Week 22.
Period: Overall Study
Arm/Group | Placebo | MEDI9929 280 mg
Started | 57 | 56
Treated | 56 | 55
Completed | 49 | 48
Not Completed | 8 | 8
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 5 | 6
Not completed — Not Treated | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent-To-Treat (ITT) population included all participants who were randomized and received any study investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | MEDI9929 280 mg | Total
Number analyzed (Participants) | 56 | 55 | 111
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.8 (15.3) | 38.5 (14.9) | 38.7 (15.0)
Age, Customized [Count of Participants; unit: Participants]
  18-35 years | 28 | 27 | 55
  36-75 years | 28 | 28 | 56
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 23 | 49
  Male | 30 | 32 | 62
Eczema Area and Severity Index Score [Count of Participants; unit: Participants] — The eczema area and severity index (EASI) evaluates 4 natural anatomical regions for severity (0 [none] to 3 [severe]) and extent of key disease signs and focuses on the key acute and chronic signs of inflammation (erythema, induration/papulation, excoriation, and lichenification). The total score is the sum of the four body-region scores, maximum=72, minimum=0. The higher values indicating more severe disease.
  Participants
    <= 25 points | 36 | 33 | 69
    > 25 points | 20 | 22 | 42
Investigator's Global Assessment [Count of Participants; unit: Participants] — The investigator's global assessment (IGA) allows investigators to assess overall disease severity at one given time point and consists of a 5-point severity scale from clear to severe disease (0 = clear, 1 = almost clear, 2 = mild disease, 3 = moderate disease, and 4 = severe disease).
  Participants
    Category 2 | 0 | 1 | 1
    Category 3 | 46 | 44 | 90
    Category 4 | 10 | 10 | 20
Atopic Dermatitis Status [Count of Participants; unit: Participants]
  IgE >= 150 kU/L and Positive Serum Specific IgEa | 50 | 47 | 97
  IgE >= 150 kU/L and Negative Serum Specific IgE | 2 | 0 | 2
  IgE < 150 kU/L and Positive Serum Specific IgE | 3 | 3 | 6
  IgE < 150 kU/L and Negative Serum Specific IgEb | 1 | 3 | 4
  Missing | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Greater Than or Equal to (>=) 50 Percent (%) Reduction From Baseline in Eczema Area and Severity Index (EASI 50) at Week 12
Description: The eczema area and severity index (EASI) evaluates 4 natural anatomical regions for severity (0 [none] to 3 [severe]) and extent of key disease signs and focuses on the key acute and chronic signs of inflammation (erythema, induration/papulation, excoriation, and lichenification). The total score is the sum of the four body-region scores, maximum=72, minimum=0. The higher values indicating more severe disease. The EASI50 responder defined as a participant who achieved at least 50% reduction in EASI score from baseline.
Time Frame: Baseline (Day 1) and Week 12
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | MEDI9929 280 mg
Number analyzed (Participants) | 56 | 55
Percentage of participants | 48.2 | 64.7
Statistical Analysis 1: Comparison: Placebo vs MEDI9929 280 mg; Test type: Superiority; Odds Ratio (OR) = 1.97, 95% CI 2-sided [0.90 to 4.33]

2. Secondary Outcome: Percentage of Participants Achieving >= 75 % Reduction From Baseline in EASI75 at Week 12
Description: The EASI evaluates 4 natural anatomical regions for severity (0 [none] to 3 [severe]) and extent of key disease signs and focuses on the key acute and chronic signs of inflammation (erythema, induration/papulation, excoriation, and lichenification). The total score is the sum of the four body-region scores, maximum=72, minimum=0. The higher values indicating more severe disease. The EASI75 responder defined as a participant who achieves at least a 75% reduction in EASI score from baseline.
Time Frame: Baseline (Day 1) and Week 12
Population: ITT population included all participants who were randomized and received any study investigational product.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | MEDI9929 280 mg
Number analyzed (Participants) | 56 | 55
Percentage of participants | 19.8 | 24.4

3. Secondary Outcome: Mean Change From Baseline in EASI Total Score at Week 12
Description: The EASI evaluates 4 natural anatomical regions for severity (0 [none] to 3 [severe]) and extent of key disease signs and focuses on the key acute and chronic signs of inflammation (erythema, induration/papulation, excoriation, and lichenification). The total score is the sum of the four body-region scores, maximum=72, minimum=0. The higher values indicating more severe disease.
Time Frame: Baseline (Day 1) and Week 12
Population: ITT population included all participants who were randomized and received any study investigational product.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | MEDI9929 280 mg
Number analyzed (Participants) | 56 | 55
units on a scale
  Baseline | 24.48 (11.21) | 24.05 (12.38)
  Week 12: number analyzed (Participants) | 50 | 49
  Week 12 | -11.23 (8.73) | -12.16 (9.96)

4. Secondary Outcome: Percentage of Participants Achieving Investigator's Global Assessment (IGA) Response of 0 (Clear) or 1 (Almost Clear) and at Least a 2-Grade Reduction From Baseline
Description: The investigator's global assessment (IGA) allows investigators to assess overall disease severity at one given time point and consists of a 5-point severity scale from clear to severe disease (0 = clear, 1 = almost clear, 2 = mild disease, 3 = moderate disease, and 4 = severe disease). A participant has IGA response if they achieve a score of 0 (clear) or 1 (almost clear) and at least a 2-grade reduction from baseline.
Time Frame: Baseline (Day 1) and Week 12
Population: ITT population included all participants who were randomized and received any study investigational product.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | MEDI9929 280 mg
Number analyzed (Participants) | 56 | 55
Percentage of participants | 12.8 | 19.3

5. Secondary Outcome: Mean Change From Baseline in the Scoring of Atopic Dermatitis (SCORAD) at Week 12
Description: The scoring of atopic dermatitis (SCORAD) is a clinical tool for assessing the severity (that is, extent, intensity) of atopic dermatitis (AD). The tool evaluates the extent and intensity of the AD lesions, along with participant symptoms. The range of the SCORAD is 0-103, where 0 indicates no eczema. The higher values indicating more severe disease.
Time Frame: Baseline (Day 1) and Week 12
Population: ITT population included all participants who were randomized and received any study investigational product.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | MEDI9929 280 mg
Number analyzed (Participants) | 56 | 55
units on a scale
  Baseline | 58.66 (13.32) | 57.68 (14.80)
  Week 12: number analyzed (Participants) | 50 | 49
  Week 12 | -19.35 (17.49) | -24.24 (16.94)

6. Secondary Outcome: Percentage of Participants Achieving >= 50% Reduction From Baseline in SCORAD 50
Description: The SCORAD is a clinical tool for assessing the severity (that is, extent, intensity) of atopic dermatitis (AD). The tool evaluates the extent and intensity of the AD lesions, along with participant symptoms. The range of the SCORAD is 0-103, where 0 indicates no eczema. The higher values indicating more severe disease. The SCORAD 50 responder defined as a participant who achieves at least a 50% reduction in SCORAD score from baseline.
Time Frame: Baseline (Day 1) and Week 12
Population: ITT population included all participants who were randomized and received any study investigational product.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | MEDI9929 280 mg
Number analyzed (Participants) | 56 | 55
Percentage of participants | 29.4 | 41.0

7. Secondary Outcome: Percentage of Participants Achieving >= 75% Reduction From Baseline in SCORAD 75
Description: The SCORAD is a clinical tool for assessing the severity (that is, extent, intensity) of atopic dermatitis (AD). The tool evaluates the extent and intensity of the AD lesions, along with participant symptoms. The range of the SCORAD is 0-103, where 0 indicates no eczema. The higher values indicating more severe disease. The SCORAD 75 responder is defined as a participant who achieves at least a 75% reduction in SCORAD score from baseline.
Time Frame: Baseline (Day 1) and Week 12
Population: ITT population included all participants who were randomized and received any study investigational product.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | MEDI9929 280 mg
Number analyzed (Participants) | 56 | 55
Percentage of participants | 7.4 | 9.8

8. Secondary Outcome: Mean Change From Baseline in Average Pruritus Numeric Rating Scale (NRS) at Week 12
Description: Pruritus is assessed using an Numeric Rating Scale (NRS) (0 - 10) with 0= no itch and 10= worst imaginable itch. Daily pruritus assessments were summarized as weekly peak score and a change from baseline in weekly peak score was calculated.
Time Frame: Baseline (Day 1) and Week 12
Population: ITT population included all participants who were randomized and received any study investigational product.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | MEDI9929 280 mg
Number analyzed (Participants) | 56 | 55
units on a scale
  Baseline: number analyzed (Participants) | 55 | 55
  Baseline | 5.15 (2.10) | 5.26 (2.02)
  Week 12: number analyzed (Participants) | 48 | 47
  Week 12 | -1.39 (1.93) | -1.90 (1.99)

9. Secondary Outcome: Mean Change From Baseline in 5-D Pruritus Score at Week 12
Description: The 5-D pruritus scale is a brief questionnaire designed to assess itch. This scale takes into account the multidimensional nature of pruritus, its impact on quality of life, and is capable of detecting change over time. The 5-D pruritus scale included 5 domains (duration, degree, direction, disability, and distribution of pruritus). The total 5-D score was obtained by scoring each of the domains separately and then summing them together. 5-D total scores ranged between 5 (no pruritus) and 25 (most severe pruritus). The higher values indicating more severe pruritus.
Time Frame: Baseline (Day 1) and Week 12
Population: ITT population included all participants who were randomized and received any study investigational product.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | MEDI9929 280 mg
Number analyzed (Participants) | 56 | 55
units on a scale
  Baseline: number analyzed (Participants) | 52 | 50
  Baseline | 16.7 (3.7) | 16.0 (3.7)
  Week 12: number analyzed (Participants) | 47 | 46
  Week 12 | -3.9 (4.5) | -3.6 (4.4)

10. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An Adverse event is any unfavourable and unintended signs (including abnormal laboratory findings), symptoms, or diseases temporally associated with use of investigational product, whether or not considered related to investigational product. Serious adverse event is any AE that resulted in:death;inpatient hospitalization or prolongation of existing hospitalization;persistent or significant disability or incapacity;is life-threatening;is a congenital anomaly/birth defect in offspring of a study participant;or was an important medical event that may not have resulted in death, threatened life,or required hospitalization and that, based on appropriate medical judgment, may have jeopardized participant and may have required medical or surgical intervention to prevent one of outcomes above. TEAEs are defined as AEs present at baseline that worsened in intensity after administration of study drug, or events absent at baseline that emerged after administration of study drug until Week 22.
Time Frame: From treatment administration (Day1) to 22 weeks
Population: As-treated population included all participants who received any study drug. Participants who received at least one dose of MEDI9929 during study, regardless of randomized treatment assignment, were analyzed under MEDI9929. One participant who randomized to placebo but received an incorrect first dose of MEDI9929 was included in "MEDI9929" group.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI9929 280 mg
Number analyzed (Participants) | 55 | 56
Participants
  TEAEs | 40 | 38
  TESAEs | 3 | 2

11. Secondary Outcome: Mean Trough Serum Concentration of MEDI9929
Description: The mean serum concentrations of MEDI9929 was observed at specified timepoints.
Time Frame: Week 0 (Pre dose), Weeks 4, 8, and 12 (post dose)
Population: PK population included all participants who received MEDI9929 and had a sufficient number of serum concentration measurements for computing PK parameters.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | MEDI9929 280 mg
Number analyzed (Participants) | 55
mcg/mL
  Week 0: number analyzed (Participants) | 50
  Week 0 | NA (NA) — All pre-first-dose values were below the limit of quantification and not calculated.
  Week 4: number analyzed (Participants) | 50
  Week 4 | 34.7 (10.9)
  Week 8: number analyzed (Participants) | 48
  Week 8 | 50.5 (17.5)
  Week 12: number analyzed (Participants) | 50
  Week 12 | 54.9 (21.5)

12. Secondary Outcome: Number of Participants Who Developed Detectable MEDI9929 Anti-drug Antibodies
Description: A participant was considered ADA-positive across the study if they had a positive reading (titer of 50 or higher) at any time point during the study period.
Time Frame: Baseline (Day 1) to Week 22
Population: ITT population included all participants who were randomized and received any study investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI9929 280 mg
Number analyzed (Participants) | 56 | 55
Participants
  Baseline | 2 | 1
  Week 22: number analyzed (Participants) | 47 | 48
  Week 22 | 2 | 0

ADVERSE EVENTS:
Time Frame: From treatment administration (Day1) to 22 weeks
Description: AEs were reported for As-treated population, which included all participants who received any study drug. Participants who received at least one dose of MEDI9929, regardless of randomized treatment, were analyzed under MEDI9929. One participant who randomized to placebo but received an incorrect first dose of MEDI9929 was included in MEDI9929 group
Arm/Group | Placebo | MEDI9929 280 mg
Serious Adverse Events (participants affected / at risk) | 3/55 | 2/56
Other Adverse Events (participants affected / at risk) | 33/55 | 29/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=55) | MEDI9929 280 mg (N=56)
Chest pain (General disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Infected dermal cyst (Infections and infestations) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=55) | MEDI9929 280 mg (N=56)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 5 (6)
Influenza like illness (General disorders) | 0 (0) | 2 (2)
Injection site erythema (General disorders) | 0 (0) | 3 (3)
Food allergy (Immune system disorders) | 0 (0) | 2 (2)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 11 (14) | 13 (15)
Sinusitis (Infections and infestations) | 2 (2) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 7 (8) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 3 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 7 (9) | 5 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises on-going studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.